CLINICAL TRIAL: NCT01034696
Title: Pain Prevalence and Risk Factors Amongst Sarcoma/Melanoma Oncology Outpatients. A Baseline, Cross Sectional Study Towards a Pain Free Hospital
Brief Title: Pain Prevalence and Risk Factors Among Sarcoma/Melanoma Oncology Patients in an Outpatients Setting
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr John Williams, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR3224
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma; Melanoma
MeSH Terms: conditions — Sarcoma; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this research project is to estimate the number of patients with sarcoma or melanoma attending an outpatients clinic that are in pain or have unmet pain needs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoma or melanoma cancer
* Able to respond to an assessment in written English.
* Able to provide informed consent to participate in the study.

Exclusion Criteria:

* Patients whose health would be compromised by participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants attending sarcoma and melanoma out patients clinics at the Royal Marsden Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with significant pain and the proportion of patients with a negative score on the pain management index (PMI)

SECONDARY OUTCOMES:
Proportion of patients with neuropathic pain.
Potential predictors of pain. The variables tested as potential risk factors will be age, tumour type, gender and treatment type.
We will also seek to identify potential predictors of pain intensity in patients that do have pain. In addition to the risk factors already mentioned above, duration and cause of pain will also be tested in this case as potential pain predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Dr John Williams, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom